CLINICAL TRIAL: NCT05975944
Title: A Phase Ib/II Clinical Study Evaluating the Safety, Tolerability, and Efficacy of Selinexor Combined With Olaparib in the Treatment of Recurrent/Refractory Extensive-stage Small Cell Lung Cancer
Brief Title: Study of Selinexor Combined With Olaparib in Relapsed/Refractory Extensive Stage Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOS-001
Record Dates: First submitted 2023-05-28; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-05

CONDITIONS: Extensive-stage Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dose-escalation part of phase Ib clinical trial (Experimental): Dose level 1: Selinexor 40mg PO QW, Olaparib 150mg PO BID; Dose level 2: Selinexor 60mg PO QW, Olaparib 150mg PO BID; Dose level 3: Selinexor 80mg PO QW, Olaparib 150mg PO BID.
  Interventions: Drug: Selinexor，Olaparib

INTERVENTIONS:
Drug: Selinexor，Olaparib — Dose level 1: Selinexor 40mg PO QW, Olaparib 150mg PO BID; Dose level 2: Selinexor 60mg PO QW, Olaparib 150mg PO BID; Dose level 3: Selinexor 80mg PO QW, Olaparib 150mg PO BID.

SUMMARY:
This study is a multicenter, single arm, open, non-randomized, dose-escalation/ expansion phase Ib/II clinical study. The dose-escalation part of phase Ib clinical trial was conducted according to the Bayesian Optimal Interval Design (BOIN), with a total of three dose groups: low, medium, and high. Dose level 1: Selinexor 40mg PO QW, Olaparib 150mg PO BID; Dose level 2: Selinexor 60mg PO QW, Olaparib 150mg PO BID; Dose level 3: Selinexor 80mg PO QW, Olaparib 150mg PO BID. The number of patients in each group is 3, with a maximum sample size of 9, to evaluate the safety and effectiveness of the medication, and to provide a basis for recommended phase II dose (RP2D). Eligible subjects received medication on the first day and then entered a 21 day observation period of dose-limiting toxicity (DLT). DLT is defined as the occurrence of level 3 non hematological toxicity or level 4 hematological toxicity. Evaluate the efficacy every 6 weeks. In this study, an independent Data Safety Monitoring Committee (DSMC) and an Independent Review Committee (IRC) were established to regularly review the safety and effectiveness data of each research center, with the aim of protecting subjects safety, ensuring the reliability of clinical trials and the objectivity of trial results.

DETAILED DESCRIPTION:
This study is a multicenter, single arm, open, non-randomized, dose-escalation/ expansion phase Ib/II clinical study. The dose-escalation part of phase Ib clinical trial was conducted according to the Bayesian Optimal Interval Design (BOIN), with a total of three dose groups: low, medium, and high. Dose level 1: Selinexor 40mg PO QW, Olaparib 150mg PO BID; Dose level 2: Selinexor 60mg PO QW, Olaparib 150mg PO BID; Dose level 3: Selinexor 80mg PO QW, Olaparib 150mg PO BID. The number of patients in each group is 3, with a maximum sample size of 9, to evaluate the safety and effectiveness of the medication, and to provide a basis for recommended phase II dose (RP2D). Eligible subjects received medication on the first day and then entered a 21 day observation period of dose-limiting toxicity (DLT). DLT is defined as the occurrence of level 3 non hematological toxicity or level 4 hematological toxicity. Evaluate the efficacy every 6 weeks. In this study, an independent Data Safety Monitoring Committee (DSMC) and an Independent Review Committee (IRC) were established to regularly review the safety and effectiveness data of each research center, with the aim of protecting subjects safety, ensuring the reliability of clinical trials and the objectivity of trial results.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of SCLC is confirmed by histology or cytology, and according to VALSG and AJCC8, the imaging diagnosis is extensive stage.
* The condition progresses after receiving at least 1 line of treatment, and within 6 months after the last treatment.
* The expected survival time is not less than 12 weeks.
* According to RECIST V1.1, there is at least one measurable lesion that has not undergone radiation therapy.
* The Eastern Cooperative Oncology Group (ECOG) physical condition score is evaluated as 0 or 1.
* When screening, there is sufficient bone marrow reserve, and no blood transfusion or hematopoietic stimulating factor treatment has been received 10 days before the test. The definition is as follows: absolute neutrophil counts (ANC) ≥ 1.5×109/L, platelet (PLT) ≥ 100×109/L and hemoglobin (HGB) ≥ 90g/L.
* Appropriate organ function during screening, meeting the following criteria: aspartate aminotransferase (AST) ≤ 2.5×ULN (with liver metastasis ≤ 5×ULN); alanine aminotransferase (ALT) ≤ 2.5ULN (with liver metastasis ≤ 5ULN); total serum bilirubin ≤ 1.5×ULN (with tumor infiltration ≤ 3×ULN); serum creatinine (Scr) ≤ 1.5×ULN, or creatinine clearance rate ≥ 60mL/min; international normalized ratio (INR) ≤ 1.5×ULN, and activated partial thromboplastin time (APTT) ≤ 1.5×ULN; the urine pregnancy test for women of childbearing age needs to be negative, and any male and female patients with fertility must agree to use effective contraceptive methods throughout the entire study process and for at least 1 year after treatment.

Exclusion Criteria:

* During screening, patients with symptomatic central nervous system (CNS) metastasis (asymptomatic CNS metastasis, or asymptomatic and stable condition after local treatment for 4 weeks can be enrolled).
* Individuals with a history of central nervous system diseases before screening, such as epilepsy, cerebral ischemia/bleeding, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, mental illness, or any autoimmune disease associated with central nervous system involvement.
* Received chemotherapy, radiation therapy, immunotherapy, targeted therapy, biological therapy, endocrine therapy within 4 weeks of screening, and was evaluated by the researcher as not suitable for enrollment.
* The adverse reactions of previous anti-tumor treatments have not yet recovered to level 1 (CTCAE5.0), except for toxicity that the researchers have determined to have no safety risk, such as hair loss and level 2 peripheral neurotoxicity.
* Those who discontinue systemic hormone therapy for less than 72 hours before the first administration, but are allowed to use physiological replacement doses of hormones (such as prednisone < 10mg/d or equivalent).
* Received organ/tissue transplantation before screening.
* Prior to screening, it was known that the patient had active systemic autoimmune diseases and was currently undergoing treatment.
* Those who meet any of the following conditions during screening: hepatitis B surface antigen (HBsAg) is positive, and the copy number of HBV DNA is greater than the measurable lower limit; hepatitis C antibody (HCV Ab) is positive; treponema pallidum antibody (TP-Ab) is positive; HIV antibody is positive; The copy numbers of EBV-DNA and CMV-DNA are higher than the measurable lower limit.
* Individuals who have undergone major surgery or experienced significant trauma within 4 weeks prior to screening, or who require elective surgery during the trial period, have been evaluated by the researchers as unsuitable for inclusion.
* Within 2 years prior to screening or currently suffering from other malignant tumors.
* When screening, the heart meets any of the following conditions: New York Heart Association (NYHA) ≥ Level II, Left Ventricular Ejection Fraction (LVEF) ≤ 50% (ECHO); Hypertension (systolic blood pressure ≥ 140mmHg and/or diastolic blood pressure ≥ 90mmHg) or pulmonary hypertension that has not been controlled after standardized treatment; Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other Grade 3 or higher cardiovascular and cerebrovascular events occurred within 6 months before the first administration; valvular disease with clinical significance; There are serious cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias that require clinical intervention, II-III degree atrioventricular block, etc.
* Patients with tumor involving the atrium or ventricle during screening.
* When screening, there are clinical emergencies that require urgent treatment due to tumor obstruction or compression (such as intestinal obstruction or vascular compression).
* Individuals with active bleeding during screening.
* Those with a history of deep vein thrombosis or pulmonary embolism within 6 months before screening.
* Individuals who have received live vaccines within 6 weeks before screening.
* Subjects with uncontrolled systemic bacterial, viral, or fungal infections after optimal treatment.
* Participated in other interventional clinical studies within 4 weeks before the first administration.
* Individuals with poor adherence or those who are deemed unsuitable for clinical trials by researchers due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
MTD | through study completion, an average of 1 year
  MTD
ORR | through study completion, an average of 1 year
  ORR

SECONDARY OUTCOMES:
DCR | through study completion, an average of 1 year
  DCR
PFS | through study completion, an average of 1 year
  PFS
OS | through study completion, an average of 1 year
  OS

CONTACTS AND LOCATIONS:
Overall Officials: huang ding zhi, M.D., Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individul participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be reviewed by an external indepentent Review Panel. Requesdtors will be required to sign a Data Access Agreement.
URL: http://www.cttq.com/

REFERENCES:
- [Result] Wang J, Sun T, Meng Z, Wang L, Li M, Chen J, Qin T, Yu J, Zhang M, Bie Z, Dong Z, Jiang X, Lin L, Zhang C, Liu Z, Jiang R, Yang G, Li L, Zhang Y, Huang D. XPO1 inhibition synergizes with PARP1 inhibition in small cell lung cancer by targeting nuclear transport of FOXO3a. Cancer Lett. 2021 Apr 10;503:197-212. doi: 10.1016/j.canlet.2021.01.008. Epub 2021 Jan 23. PMID 33493586